CLINICAL TRIAL: NCT02417519
Title: Acute Effects of Light and Dark Roasted Coffee on Glucose Tolerance: A Randomized, Controlled Crossover Trial in Healthy Volunteers
Brief Title: Coffee Roasting and Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: M217
Record Dates: First submitted 2015-04-11; First posted 2015-04-15 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Oral Glucose Tolerance
Keywords: Coffee; Chlorogenic acid; Insulin; Appetite; Metabolomics
MeSH Terms: conditions — Insulin Resistance | interventions — Coffee; Glucose Tolerance Test; Water

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence A (Experimental): The meal study was performed with dark roast coffee (DAR), light roast coffe (LIR), or water (CTR) in a random sequence. Sequance A was DAR-LIR-CTR
  Interventions: Other: DAR; Other: LIR; Other: CTR
- Sequence B (Experimental): The meal study was performed with dark roast coffee (DAR), light roast coffe (LIR), or water (CTR) in a random sequence. Sequance B was DAR-CTR-LIR
  Interventions: Other: DAR; Other: LIR; Other: CTR
- Sequance C (Experimental): The meal study was performed with dark roast coffee (DAR), light roast coffe (LIR), or water (CTR) in a random sequence. Sequance C was LIR-DAR-CTR
  Interventions: Other: DAR; Other: LIR; Other: CTR
- Sequence D (Experimental): The meal study was performed with dark roast coffee (DAR), light roast coffe (LIR), or water (CTR) in a random sequence. Sequance D was LIR-CTR-DAR
  Interventions: Other: DAR; Other: LIR; Other: CTR
- Sequence E (Experimental): The meal study was performed with dark roast coffee (DAR), light roast coffe (LIR), or water (CTR) in a random sequence. Sequance E was CTR-DAR-LIR
  Interventions: Other: DAR; Other: LIR; Other: CTR
- Sequence F (Experimental): The meal study was performed with dark roast coffee (DAR), light roast coffe (LIR), or water (CTR) in a random sequence. Sequance F was CTR-LIR-DAR
  Interventions: Other: DAR; Other: LIR; Other: CTR

INTERVENTIONS:
Other: DAR — Volunteers ingested 300 mL of coffee with a dark roast containing low levels of chlorogenic acids followed 30 min later by by 75g glucose and 300 mL water
  Other Names: 300 mL of coffee with a dark roast + OGTT
Other: LIR — Volunteers ingested 300 mL of coffee with a light roast containing high levels of chlorogenic acids followed 30 min later by by 75g glucose and 300 mL water
  Other Names: 300 mL of coffee with a light roast + OGTT
Other: CTR — Volunteers ingested 300 mL of water containing no chlorogenic acids followed 30 min later by by 75g glucose and 300 mL water
  Other Names: 300 mL of water + OGTT

SUMMARY:
Chlorogenic acid (CGA) in coffee may lower the postprandial glucose response. CGA is destroyed by dark roasting. In a controlled crossover trial, 11 healthy fasted volunteers consumed 300 mL of either light (LIR) or dark (DAR) roasted coffee, or water, followed 30 min later by a 75-g oral glucose tolerance test (OGTT). Plasma glukose and insulin, appetite, and plasma and urine metabolic profiles will be analysed. The primary aim is to investigate whether roasting affects the postprandial glucose area under the curve (AUC).

DETAILED DESCRIPTION:
Epidemiologic evidence suggests that coffee consumption is associated with a lower risk of type 2 diabetes. Coffee contains caffeine and several other components that may modulate glucose regulation. The chlorogenic acids (CGA) in coffee have been indicated as constituents that may help to normalize the acute glucose response after a carbohydrate challenge. The aim of this study was to investigate whether two coffee beverages that differ in CGA content due to different roasting degrees will affect glucose regulation differently.

In a controlled crossover trial, 11 healthy fasted volunteers consumed 300 mL of either light roasted (LIR) or dark roasted (DAR) coffee, or water, followed 30 min later by a 75-g oral glucose tolerance test (OGTT). Blood samples were drawn at baseline, 30, 60 and 120 min. Differences in glucose and insulin responses and insulin sensitivity index (ISI) were analyzed. The CGA and caffeine contents in the coffees were analyzed using UPLC-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

Body mass index (BMI) of 18.0-30.0 kg/m2 and with no known diseases

Exclusion Criteria:

* systemic infections,
* psychiatric or metabolic disorders,
* known food allergies or intolerances related to the products used in the study (e.g. dairy or gluten),
* ongoing or former drug abuse,
* high intake of alcohol (defined as a weekly intake of >7 units for women and > 14 units for men),
* pregnancy or ongoing planning of pregnancy,
* vegetarianism or veganism,
* participation in other scientific studies during the study period, and
* blood donation during - or in the month leading up to - the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Plasma glucose Area Under the Curve (Glucose AUC) | 0-120 min
  The area under the plasma glucose concentration curve was calculated from 0-120min after 75g glucose was ingested.

SECONDARY OUTCOMES:
Plasma glucose concentrations | 30, 60 and120 min
  changes in the glucose concentration determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate.
Serum Insulin Area Under the Curve | 0-120 min
  Area under the curve (AUC) for serum insulin
Serum insulin concentrations | 30, 60 and120 min
  changes in the insulin concentration determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate.
ISI(0-120) | 0-120min
  Matsuda's Insulin sensitivity index
Metabolic profile in plasma | 0-24 hours
  Metabolic profile of plasma measured in all samples collected before the meal and postprandially from 0-120 min as well as in samples collected up to 24 hrs later.
Metabolic profile in urine | 0-24 hours
  Metabolic profile of urine samples measured in all samples collected before the meal and postprandially from 0-120 min 120-240min as well as in samples collected up to 24 hrs later.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark